CLINICAL TRIAL: NCT00636337
Title: TRICCS: Targeting Inattention in Childhood Cancer Survivors
Brief Title: Inattention in Childhood Cancer Survivors
Acronym: TRICCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00003249; NCT00735202 (obsolete NCT alias)
Record Dates: First submitted 2008-02-28; First posted 2008-03-14 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Childhood Cancer
Keywords: Pediatric; Brain Tumor; Acute Lymphoblastic Leukemia; Inattention; Childhood cancer survivors
MeSH Terms: conditions — Neoplasms; Brain Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants meeting inclusion criteria will be provided with a laptop computer outfitted with a wireless card for the duration of the intervention and will be trained in the use of RoboMemo in the clinic by study personnel. Although many participants may have ready access to home computers, we decided that all participants will be required to use laptops provided by the study for two reasons: 1) to ensure that coaches and participants are blind to treatment condition (as described above), and 2) to ensure that participants will always have access to the intervention program (i.e., they will not compete with other family members for computer time). Once trained, children will complete the intervention at home. The intervention will consist of four 30- to 45-minute sessions per week for 8 weeks (total = 32 sessions). This intervention schedule is similar to the schedule employed by Klingberg and colleagues in their home-based CT trials with ADHD children.
  Interventions: Behavioral: Attention Training
- 2 (Placebo Comparator): The design will be a double-blind, placebo-controlled trial in which half of the participants will be randomized to the intervention condition and half will receive a comparison computer program. Specifically, participants assigned to the comparison (placebo) condition will complete a modified version of the CT at home. The treatment and comparison CT programs begin identically, at the lowest difficulty level. Those in the treatment condition will complete activities of increasing difficulty over the intervention period. Those in the placebo condition, in contrast, will complete the same basic tasks during each session of the intervention, regardless of performance. In this way, a true estimate can be obtained of the efficacy of the treatment program.
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Attention Training — Computer program training for attention difficulties.
  Other Names: TRICCS; RoboMemo
  Arms: 1
Behavioral: Placebo — Comparison computer program
  Arms: 2

SUMMARY:
Specific Aim 1: To assess the feasibility and acceptability of a home-based, computerized cognitive training program with survivors of central nervous system-impacting pediatric cancer (e.g. acute lymphoblastic leukemia, brain tumors).

Specific Aim 2: To estimate the effect size of this cognitive training program on measures of attention and working memory in survivors of childhood cancer in order to determine whether a larger-scale clinical trial is warranted.

DETAILED DESCRIPTION:
After obtaining written informed consent (parent) and assent (child), screening procedures will include administration of an abbreviated intellectual test battery, a working memory battery, and a computerized attention measure to the survivor (see specific Measures below). Our goal is to enroll 24 (12 ALL, 12 brain tumor) participants in the intervention phase of this prospective pilot study. To reach this goal, we anticipate needing to screen approximately 50 survivors, though enrollment will end when, or continue until, 24 eligible participants are identified and randomized to the intervention phase. Parents will complete questionnaire measures regarding their child's adaptive, behavioral, emotional, and attentional functioning. Follow-up interviewing will be conducted to clarify any potential problems identified on the questionnaires. The entire screening procedure is estimated to take approximately 90 minutes for the survivor and 30-45 minutes for parents. To maximize efficiency, two study personnel will work with families - one will complete testing with the child, while the other will complete questionnaires and follow-up interviewing with the parent. The design will be a double-blind, placebo-controlled trial in which half of the participants will be randomized to the intervention condition and half will receive a comparison computer program. Specifically, participants assigned to the comparison (placebo) condition will complete a modified version of the CT at home. The treatment and comparison CT programs begin identically, at the lowest difficulty level. Those in the treatment condition will complete activities of increasing difficulty over the intervention period. Those in the placebo condition, in contrast, will complete the same basic tasks during each session of the intervention, regardless of performance. In this way, a true estimate can be obtained of the efficacy of the treatment program.

ELIGIBILITY:
Inclusion Criteria:

1. A T-score greater than the 75th percentile on either the Cognitive Problems/Inattention or the DSM-IV Inattention subscales of the Conners' Parent Rating Scale
2. One or more standard deviations below the mean on the Attention or Working Memory Indices of the WRAML 2 [56] or Attention or Working Memory Indices that are one or more standard deviations below the participant's estimated IQ. These criteria are similar to those used in a trial of methylphenidate with survivors of childhood cancer.

Exclusion Criteria:

1. Estimated IQ ≤ 70
2. A motor, visual, or auditory handicap that prevents computer use
3. A diagnosis of Attention-Deficit Hyperactivity Disorder (ADHD), Oppositional Defiant Disorder, depression, autism, or Pervasive Developmental Disorder
4. Insufficient fluency in English. Participants who are currently taking stimulant medications (stable dose for at least 30 days) for attentional difficulties, but who meet inclusion criteria listed below will be allowed to participate.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Memory | 2 months and 3 months

SECONDARY OUTCOMES:
Feasibility | once a month for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Hardy, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center Preston Robert Tisch Brain Tumor Center, Durham, North Carolina, United States